CLINICAL TRIAL: NCT00621231
Title: Effect of Normal Versus High Amounts of Protein Intake on Physiological Functions and Proteomics in Healthy Men
Brief Title: The Protein (Meat) and Function Study
Acronym: ProF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Model: Parallel | Purpose: Basic Science
Other Study IDs: K101
Record Dates: First submitted 2008-02-12; First posted 2008-02-22 (Estimated); Last update posted 2008-02-22 (Estimated); Status verified 2007-05

CONDITIONS: Healthy
Keywords: Protein Function; normal versus high protein intake
MeSH Terms: interventions — Proteins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- 2 (Experimental)
  Interventions: Dietary Supplement: Protein

INTERVENTIONS:
Dietary Supplement: Placebo — Placebo
  Arms: 1
Dietary Supplement: Protein — 30 E% from protein
  Arms: 2

SUMMARY:
The aim of the proposed study is to investigate the effects of different amounts of protein intake primarily from meat on muscle function, immune response, mental function, proteomics, biochemical regulators of protein metabolism, energy expenditure, and composition in young healthy males.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males, 19-40 y/o

Exclusion Criteria:

* Smokers

Ages: 19 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2007-09; Primary Completion 2007-12 (Actual); Study Completion 2008-04

CONTACTS AND LOCATIONS:
Locations (1):
- Department of human nutrition, Copenhagen, DK-Frederiksberg C, Denmark

REFERENCES:
- [Derived] Jakobsen LH, Kondrup J, Zellner M, Tetens I, Roth E. Effect of a high protein meat diet on muscle and cognitive functions: a randomised controlled dietary intervention trial in healthy men. Clin Nutr. 2011 Jun;30(3):303-11. doi: 10.1016/j.clnu.2010.12.010. Epub 2011 Jan 15. PMID 21239090